CLINICAL TRIAL: NCT01434485
Title: Nexium Capsules Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961HC00010
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Gastric Ulcer, Duodenal Ulcer, Anastomotic Ulcer, Reflux Oesophagitis,"Non-erosive Reflux Disease, Zollinger-Ellison Syndrome
Keywords: gastric ulcer, duodenal ulcer, anastomotic ulcer, reflux oesophagitis, non-erosive reflux disease, Zollinger-Ellison syndrome, Nexium
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Zollinger-Ellison Syndrome; Esophagitis, Peptic; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nexium

SUMMARY:
The purpose of this study is to confirm the safety profile / factors which impact safety and efficacy of Nexium capsules in daily clinical usage for the patients who have been prescribed Nexium for "gastric ulcer", "duodenal ulcer", "anastomotic ulcer", "reflux oesophagitis", "non-erosive reflux disease", or "Zollinger-Ellison syndrome"

DETAILED DESCRIPTION:
Nexium capsules Clinical Experience Investigation

ELIGIBILITY:
Inclusion Criteria: - Patients treated with Nexium for the first time due to gastric ulcer, duodenal ulcer, anastomotic ulcer, reflux oesophagitis, non-erosive reflux disease, Zollinger-Ellison syndrome. Exclusion Criteria: - None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Nexium for the first time due to gastric ulcer, duodenal ulcer, anastomotic ulcer, reflux oesophagitis, non-erosive reflux disease, Zollinger-Ellison syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 3691 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Drug Reactions | Patients with gastric ulcer, anastomotic ulcer or Zollinger-Ellison syndrome: 8 weeks
Number of Adverse Drug Reactions | Patients with duodenal ulcer: 6 weeks
Number of Adverse Drug Reactions | Patients with reflux oesophagitis: 8 weeks
Number of Adverse Drug Reactions | Patients with non-erosive reflux disease: 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi